CLINICAL TRIAL: NCT05019664
Title: Post-market Clinical Follow-up Study to Provide Safety, Performance and Clinical Benefits Data of the Affixus Natural Nail System Humeral Nail (Implants and Instrumentation)
Brief Title: Affixus Natural Nail System Humeral Nail PMCF
Status: Recruiting | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CMG2020-09T
Record Dates: First submitted 2021-07-06; First posted 2021-08-25 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-06

CONDITIONS: Humeral Fractures, Proximal; Humeral Fractures
MeSH Terms: conditions — Shoulder Fractures; Humeral Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: humeral fracture — Patient with either a proximal humeral fracture or humeral shaft fracture requiring surgical intervention and be eligible for fixation by intramedullary nailing.

SUMMARY:
A commercially available product clinical study which aims to confirm the safety, performance and clinical benefits to the patient of the Affixus Natural Nail upper arm (humerus) bone nail system for both the implant itself and the instrumentation used during surgery.

DETAILED DESCRIPTION:
Study objective:

The objectives of this observational, prospective study with optional retrospective enrollment are to confirm safety, performance and clinical benefits of the Affixus Natural Nail System Humeral Nail and its instrumentation by analyzing adverse event records, fracture/osteotomy healing and functional outcome and adverse events.

The safety of the system will be assessed by monitoring the frequency and incidence of adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.

The performance and clinical benefits will be evaluated by assessment of fracture/osteotomy healing and functional outcome of all enrolled study subjects.

Study Endpoints:

Primary endpoint:

The primary endpoint is bone union after 12 months since surgery.

Secondary endpoint:

The secondary endpoints will be evaluating functional outcomes (Range of Motion, & American Shoulder and Elbow Surgeons questionnaire), quality of life questionnaire (EQ-5D-5L), radiographic findings and adverse events including re-operation of all enrolled study subjects at the defined follow up time points.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older and skeletally mature.
* Patient must have either a proximal humeral fracture or humeral shaft fracture requiring surgical intervention and be eligible for fixation by intramedullary nailing.
* Patient has been or is scheduled to be treated with the Affixus Natural Nail System Humeral Nail.
* Patient must be able and willing to complete the protocol required follow-up.
* Patient must have a signed Institutional Review Board/Ethics Committee approved informed consent. (An Institutional Review Board/Ethics Committee is group that has been formally designated to review and monitor medical research involving human subjects.)
* Patients capable of understanding the surgeon's explanations and following his instructions, able and willing to participate in the follow-up program and who gave consent to take part in the study.

Exclusion Criteria:

* Distal fracture involving the olecranon fossa.
* Bone shaft having excessive bow or deformity.
* A medullary canal obliterated by a previous fracture or tumor.
* Active or previous infection.
* Skeletally immature patients.
* All concomitant diseases that can impair the functioning and the success of the implant.
* Patients with mental or neurologic conditions who are unwilling or incapable of giving proper informed consent and following postoperative care instructions.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, anticipated to be non-compliant).
* Patient known to be pregnant or breast feeding.
* Likely problems with maintaining follow-up program (e.g. patient with no fixed address, long distance, plans to move during course of study).
* Patients who have any condition that would in the judgment of the investigator place the patient at undue risk or interfere with the study.
* Not expected to survive the duration of the follow-up program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive series of 100 subjects globally implanted with the Affixus Natural Nail System Humeral Nail for temporary fixation and stabilization of fractures or osteotomies of the humerus.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-08-29 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Bone Union | 12 months
  The primary endpoint is bone union after 12 months since surgery. (Bone union defined as no pain or tenderness at the site, and strong enough to allow normal activities.)

SECONDARY OUTCOMES:
Range of Motion | 12 months
  The Range of Motion (total shoulder motion, active and passive) of the affected and contralateral (right and left) upper arm will be measured.
EQ-5D-5L | 12 months
  EQ-5D-5L Health Questionnaire is completed by the patient and assesses his/her general health status. The EQ-5D-5L is used to derive a quality of life index used for health economics considerations.
Radiographic Findings | 12 months
  Postoperative Radiographic Evaluation collects radiographic parameters like bridging callus, visible fracture line, device fracture, device loosening and union status (AP, lateral, and auxiliary view).
Adverse Events | 12 months
  Adverse Event Report is completed as needed for each complication which is noted.

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Rohmer, MSc., Study Director — Zimmer Biomet
Locations (5):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States
- UZ Leuven - Traumatology Department, Leuven, Belgium
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - General Foundation of the University of Valladolid, Valladolid
- Kantonsspital Frauenfeld, Frauenfeld, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
This aspect of the study is undecided.